CLINICAL TRIAL: NCT01339559
Title: An Open-label, Multicenter, Follow-up Study to Evaluate the Long-term Safety and Efficacy of Brivaracetam Used as Adjunctive Treatment in Subjects Aged 16 Years or Older With Epilepsy
Brief Title: Brivaracetam Safety and Efficacy Follow-up Study in Subjects With Epilepsy
Acronym: BRITE™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01379; 2010-020345-27 (EudraCT Number)
Expanded Access: NCT03532516 (Available)
Record Dates: First submitted 2011-04-19; First posted 2011-04-20 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Epilepsy
Keywords: Epilepsy; Brivaracetam; Partial Onset Seizures; Adjunctive treatment
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brivaracetam (Experimental): Brivaracetam with a maximum of 200 mg/day
  Interventions: Drug: Brivaracetam

INTERVENTIONS:
Drug: Brivaracetam — Tablet, Flexible dosing up to 200 mg/day, twice daily.
  The study will continue until either regulatory approval of brivaracetam has been granted by any Health Authority in an indication of adjunctive treatment of partial onset seizures or until the Sponsor decides to close the study, or until the investigational product development is stopped by the Sponsor.
  Other Names: UCB34714

SUMMARY:
This is a Phase 3, open label, long term follow-up (LTFU), multicenter, noncomparative, and single arm study of brivaracetam (BRV).

DETAILED DESCRIPTION:
The primary objective is to evaluate the long term safety and tolerability of BRV at individualized doses up to a maximum of 200 mg/day in epilepsy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject completed the Treatment Period of N01358 or the evaluation period of N01258
* Male/female subject from 16 years or older. Subject under 18 years may only be included where legally permitted and ethically accepted
* Subject for whom the Investigator believes a reasonable benefit from the long term administration of BRV may be expected
* Female subject without childbearing potential (premenarcheal, postmenopausal for at least 2 years, bilateral oophorectomy or tubal ligation, complete hysterectomy) are eligible

Exclusion Criteria:

* Subject has developed hypersensitivity to any components of the investigational medicinal product (IMP) or comparative drugs as stated in this protocol during the course of the core studies
* Severe medical, neurological, or psychiatric disorders, or laboratory values which may have an impact on the safety of the subject
* Poor compliance with the visit schedule or medication intake in the previous BRV study
* Planned participation in any other clinical study of another investigational drug or device during this study
* Pregnant or lactating woman
* Any medical condition which, in the Investigator's opinion, warrants exclusion
* Subject has a lifetime history of suicide attempt or has suicidal ideation in the past 6 months

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 767 (Actual)
Dates: Start 2011-05-11 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (184):
- United States (49):
  - 001, Phoenix, Arizona
  - 013, Phoenix, Arizona
  - 006, Tucson, Arizona
  - 775, Little Rock, Arkansas
  - 025, San Francisco, California
  - 060, Aurora, Colorado
  - 071, Miami, Florida
  - 027, Orlando, Florida
  - 064, Port Charlotte, Florida
  - 023, Atlanta, Georgia
  - 048, Rome, Georgia
  - 039, Boise, Idaho
  - 029, Chicago, Illinois
  - 005, Peoria, Illinois
  - 017, Winfield, Illinois
  - 020, Ames, Iowa
  - 069, Iowa City, Iowa
  - 780, Lexington, Kentucky
  - 008, Bethesda, Maryland
  - 068, Waldorf, Maryland
  - 009, Golden Valley, Minnesota
  - 032, Lebanon, New Hampshire
  - 042, Hamilton, New Jersey
  - 099, New York, New York
  - 022, New York, New York
  - 098, Poughkeepsie, New York
  - 010, Asheville, North Carolina
  - 003, Durham, North Carolina
  - 034, Cleveland, Ohio
  - 778, Columbus, Ohio
  - 070, Columbus, Ohio
  - 002, Toledo, Ohio
  - 043, Oklahoma City, Oklahoma
  - 091, Oklahoma City, Oklahoma
  - 054, Tulsa, Oklahoma
  - 015, Philadelphia, Pennsylvania
  - 028, Charleston, South Carolina
  - 021, Port Royal, South Carolina
  - 776, Nashville, Tennessee
  - 061, Austin, Texas
  - 011, Dallas, Texas
  - 777, Dallas, Texas
  - 035, Dallas, Texas
  - 049, Houston, Texas
  - 050, Mansfield, Texas
  - 036, Charlottesville, Virginia
  - 056, Spokane, Washington
  - 052, Madison, Wisconsin
  - 057, Milwaukee, Wisconsin
- Austria (3):
  - 202, Innsbruck
  - 201, Linz
  - 203, Vienna
- Belgium (2):
  - 226, Hechtel-Eksel
  - 227, Leuven
- Brazil (3):
  - 104, Belo Horizonte
  - 100, Florianópolis
  - 101, São Paulo
- Bulgaria (3):
  - 294, Blagoevgrad
  - 286, Sofia
  - 287, Sofia
- Canada (6):
  - 075, Calgary, Alberta
  - 078, London, Ontario
  - 076, Toronto, Ontario
  - 077, Greenfield Park, Quebec
  - 080, Saskatoon, Saskatchewan
  - 079, Montreal
- Czechia (8):
  - 917, Brno
  - 916, Kroměříž
  - 251, Ostrava
  - 256, Ostrava
  - 913, Ostrava Poruba
  - 252, Prague
  - 253, Prague
  - 250, Zlín
- Estonia (3):
  - 650, Tallinn
  - 652, Tallinn
  - 651, Tartu
- Finland (2):
  - 275, Kuopio
  - 276, Tampere
- France (2):
  - 301, Béthune
  - 305, Montpellier
- Germany (11):
  - 329, Berlin
  - 326, Bernau
  - 332, Bielefeld
  - 902, Erlangen
  - 331, Göttingen
  - 327, Kiel
  - 900, Marburg
  - 335, München
  - 334, Osnabrück
  - 330, Ravensburg
  - 328, Ulm
- Hong Kong (2):
  - 700, Hong Kong
  - 701, Hong Kong
- Hungary (5):
  - 410, Budapest
  - 411, Budapest
  - 412, Budapest
  - 414, Hajdú-Bihar
  - 413, Szekszárd
- India (6):
  - 731, Nashik, Maharashtra
  - 726, Bangalore
  - 727, Hyderabad
  - 729, Madurai
  - 725, Mumbai
  - 728, Mumbai
- Italy (9):
  - 378, Bari
  - 380, Florence
  - 379, Milan
  - 377, Monserrato
  - 386, Napoli
  - 376, Perugia
  - 375, Pisa
  - 383, Pozzilli
  - 384, Reggio Calabria
- Japan (5):
  - 852, Itami, Hyōgo
  - 855, Hiroshima
  - 850, Osaka
  - 851, Shizuoka
  - 854, Yokohama
- Latvia (4):
  - 627, Daugavpils
  - 629, Jēkabpils
  - 628, Riga
  - 625, Valmiera
- Lithuania (3):
  - 425, Alytus
  - 427, Kaunas
  - 426, Vilnius
- Mexico (6):
  - 126, Guadalajara, Jalisco
  - 128, Guadalajara, Jalisco
  - 129, Aguascalientes
  - 127, Culiacán
  - 125, Distrito Federal
  - 130, Mexico City
- Netherlands (3):
  - 401, Heemstede
  - 400, Heeze
  - 403, Zwolle
- Poland (15):
  - 475, Bialystok
  - 485, Gdansk
  - 791, Gdansk
  - 478, Katowice
  - 480, Katowice
  - 481, Katowice
  - 795, Katowice
  - 476, Krakow
  - 793, Krakow
  - 483, Lublin
  - 477, Poznan
  - 479, Poznan
  - 482, Poznan
  - 488, Warsaw
  - 794, Warsaw
- 038, San Juan, Puerto Rico
- Russia (6):
  - 501, Kazan'
  - 506, Kazan'
  - 502, Moscow
  - 503, Moscow
  - 509, Nizhny Novgorod
  - 508, Smolensk
- South Korea (4):
  - 753, Busan
  - 750, Seoul
  - 751, Seoul
  - 754, Seoul
- Spain (9):
  - 528, Barcelona
  - 529, Barcelona
  - 535, Barcelona
  - 540, Barcelona
  - 539, Donostia / San Sebastian
  - 532, Santiago de Compostela
  - 527, Valencia
  - 537, Valencia
  - 526, Valladolid
- Sweden (3):
  - 551, Gothenburg
  - 552, Linköping
  - 550, Stockholm
- Taiwan (4):
  - 806, Kaohsiung City
  - 801, Taichung
  - 800, Tainan
  - 803, Taoyuan District
- United Kingdom (7):
  - 602, Morriston, Swansea
  - 603, Birmingham
  - 600, London
  - 605, Middlesbrough
  - 607, Newcastle
  - 608, Salford
  - 601, Truro

REFERENCES:
- [Result] Moseley BD, Dimova S, Elmoufti S, Laloyaux C, Asadi-Pooya AA. Long-term efficacy and tolerability of adjunctive brivaracetam in adults with focal to bilateral tonic-clonic (secondary generalized) seizures: Post hoc pooled analysis. Epilepsy Res. 2021 Oct;176:106694. doi: 10.1016/j.eplepsyres.2021.106694. Epub 2021 Jun 24. PMID 34218211
- [Derived] Brandt C, Dimova S, Elmoufti S, Laloyaux C, Nondonfaz X, Klein P. Retention, efficacy, tolerability, and quality of life during long-term adjunctive brivaracetam treatment by number of lifetime antiseizure medications: A post hoc analysis of phase 3 trials in adults with focal seizures. Epilepsy Behav. 2023 Jan;138:108967. doi: 10.1016/j.yebeh.2022.108967. Epub 2022 Nov 23. PMID 36435010
- [Derived] Markham A. Brivaracetam: First Global Approval. Drugs. 2016 Mar;76(4):517-22. doi: 10.1007/s40265-016-0555-6. PMID 26899665
- [Derived] Klein P, Schiemann J, Sperling MR, Whitesides J, Liang W, Stalvey T, Brandt C, Kwan P. A randomized, double-blind, placebo-controlled, multicenter, parallel-group study to evaluate the efficacy and safety of adjunctive brivaracetam in adult patients with uncontrolled partial-onset seizures. Epilepsia. 2015 Dec;56(12):1890-8. doi: 10.1111/epi.13212. Epub 2015 Oct 16. PMID 26471380
- See also: Product Information — http://www.briviact.com/briviact-PI.pdf?v=1479491757
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in May 2011 and concluded in April 2019. 767 participants were included in the Enrolled Set but 1 participant from the United States of America was lost to follow-up and was excluded from the Safety Analysis Set.
Pre-assignment Details: Participants Flow refers to the Safety Set (SS).
Groups:
- Brivaracetam: Brivaracetam (BRV) was administered with a maximum of 200 mg/day, twice, daily, incremented by 50 mg/day on a weekly basis, during the Up-Titration. During the Down-Titration Period, the BRV dose was decreased in steps of a maximum of 50 mg/day on a weekly basis. A last down-titration step at 20 mg/day for 1 week was included prior to the Post-Treatment Period.
Period: Overall Study
Arm/Group | Brivaracetam
Started | 766
Completed | 368
Not Completed | 398
Not completed — Adverse Event | 92
Not completed — Death | 5
Not completed — Lack of Efficacy | 164
Not completed — Lost to Follow-up | 22
Not completed — Subject choice | 89
Not completed — Protocol Violation | 15
Not completed — Study closure at site | 1
Not completed — Incarcerated | 2
Not completed — Epilepsy surgery | 1
Not completed — Pregnancy planned | 2
Not completed — Left the country | 1
Not completed — Investigator decision | 2
Not completed — Patient didn't wish to continue | 1
Not completed — PI decision | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set which consisted of all participants who took at least 1 dose of study medication.
Arm/Group | Brivaracetam
Number analyzed (Participants) | 766
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19
  Between 18 and 65 years | 722
  >=65 years | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 396
  Male | 370
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 561
  African-American | 37
  Asian | 85
  Other | 77
  Missing | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Treatment-Emergent Adverse Event (TEAE)
Description: Treatment-emergent Adverse Events (TEAEs) were defined as those events which started on or after the date of first dose of investigational medicinal product (IMP), or events in which severity worsened on or after the date of first dose of study medication. The event does not necessarily have a causal relationship with that treatment or usage.
Time Frame: From Entry Visit (Month 0) until the Last Visit (up to 84 months)
Population: The Safety Set (SS) consisted of all participants who took at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Groups:
- Brivaracetam (SS): Brivaracetam (BRV) was administered with a maximum of 200 mg/day, twice, daily, incremented by 50 mg/day on a weekly basis, during the Up-Titration. During the Down-Titration Period, the BRV dose was decreased in steps of a maximum of 50 mg/day on a weekly basis. A last down-titration step at 20 mg/day for 1 week was included prior to the Post-Treatment Period. Participants formed the Safety Set (SS).
Arm/Group | Brivaracetam (SS)
Number analyzed (Participants) | 766
Percentage of participants | 83.9

2. Primary Outcome: Percentage of Participants Who Withdrew Due to Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant or trial subject that is administered a drug or biologic (medicinal product) or that is using a medical device. The event does not necessarily have a causal relationship with that treatment or usage.
Time Frame: From Entry Visit (Month 0) until the Last Visit (up to 84 months)
Population: The Safety Set (SS) consisted of all participants who took at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Brivaracetam (SS)
Number analyzed (Participants) | 766
Percentage of participants | 11.9

3. Primary Outcome: Percentage of Participants With at Least One Serious Adverse Event (SAE)
Description: A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalization or prolongation of existing hospitalization
  * Is a congenital anomaly or birth defect
  * Is as infection that requires treatment parenteral antibiotics
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients or may require medical or surgical intervention to prevent any of the above.
Time Frame: From Entry Visit (Month 0) until the Last Visit (up to 84 months)
Population: The Safety Set (SS) consisted of all participants who took at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Brivaracetam (SS)
Number analyzed (Participants) | 766
Percentage of participants | 18.4

4. Secondary Outcome: Partial Onset Seizure (POS) (Type I) Frequency Per 28 Days During the Evaluation Period
Description: The 28 day adjusted seizure frequency was calculated by dividing the number of partial seizures by the number of days for which the diary was completed, and multiplying the resulting value by 28.
Time Frame: From Baseline of the previous study until the Last Visit (up to 84 months)
Population: The Partial Onset Seizure (POS) Efficacy Analysis Set consisted of all subjects with POS who took at least 1 dose of study drug and had at least 1 seizure diary day during the Evaluation Period.
Measure: Median (Inter-Quartile Range); unit: Seizures per 28 days
Groups:
- Brivaracetam (POS Efficacy): Brivaracetam (BRV) was administered with a maximum of 200 mg/day, twice, daily, incremented by 50 mg/day on a weekly basis, during the Up-Titration. During the Down-Titration Period, the BRV dose was decreased in steps of a maximum of 50 mg/day on a weekly basis. A last down-titration step at 20 mg/day for 1 week was included prior to the Post-Treatment Period. Participants formed the Partial Onset Seizure Efficacy Set (POS Efficacy).
Arm/Group | Brivaracetam (POS Efficacy)
Number analyzed (Participants) | 749
Seizures per 28 days
  Baseline | 9.7 [5.5 to 23.7]
  On Treatment | 4.2 [1.4 to 12.7]

5. Secondary Outcome: Percent Change in Partial Onset Seizure (POS) (Type I) Frequency Per 28 Days From Baseline of the Previous Study to the Evaluation Period
Description: The percent change from the previous study baselines, in Partial Onset Seizure (POS) (Type I) frequency per 28 days is defined as:
  (the value at the previous study baselines) minus (the value at each time-points during the evaluation period) divided by the value at the previous study baselines.
  Note: Since N01258 was a safety study, participants were not required to meet seizure frequency requirements during the Baseline Period, and the Baseline Period was short (ie, 7 days). Therefore, participants from N01258 were excluded from efficacy summaries in the variable of percent change in POS frequency.
Time Frame: From Baseline of the previous study until the Last Visit (up to 84 months)
Population: The Partial Onset Seizure (POS) Efficacy Analysis Set consisted of all subjects with POS who took at least 1 dose of study drug and had at least 1 seizure diary day during the Evaluation Period.
  Participants from N01258 were excluded from this analysis.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Brivaracetam (POS Efficacy)
Number analyzed (Participants) | 675
Percent change | 52.0 [16.8 to 81.5]

6. Secondary Outcome: Responder Rate in POS (Type I) Frequency Over the Evaluation Period
Description: A responder is defined as a subject with a ≥ 50% reduction in seizure frequency from the Baseline Period of the previous study.
  Note: Since N01258 was a safety study, participants were not required to meet seizure frequency requirements during the Baseline Period, and the Baseline Period was short (ie, 7 days). Therefore, participants from N01258 were excluded from efficacy summaries in the variable of responder rates in POS frequency.
Time Frame: From Baseline of the previous study until the Last Visit (up to 84 months)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Brivaracetam (POS Efficacy)
Number analyzed (Participants) | 675
Percentage of participants | 51.7

ADVERSE EVENTS:
Time Frame: From Entry Visit (Month 0) until the Last Visit (up to 84 months)
Arm/Group | Brivaracetam (SS)
All-Cause Mortality (participants affected / at risk) | 5/766
Serious Adverse Events (participants affected / at risk) | 140/766
Other Adverse Events (participants affected / at risk) | 421/766
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivaracetam (SS) (N=766)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1)
Hypoplastic anaemia (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Sickle cell anaemia (Congenital, familial and genetic disorders) | 1 (1)
Goitre (Endocrine disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Oesophageal perforation (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Device malfunction (General disorders) | 1 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 3 (3)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5)
Sepsis (Infections and infestations) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Gastroenteritis escherichia coli (Infections and infestations) | 1 (1)
Infected cyst (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Otitis media chronic (Infections and infestations) | 1 (1)
Perineal abscess (Infections and infestations) | 1 (1)
Pharyngitis bacterial (Infections and infestations) | 1 (1)
Typhoid fever (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 3 (4)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2)
Brain contusion (Injury, poisoning and procedural complications) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 2 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Nail injury (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Skeletal injury (Injury, poisoning and procedural complications) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Diagnostic procedure (Investigations) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Troponin increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Gliomatosis cerebri (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Convulsion (Nervous system disorders) | 15 (16)
Status epilepticus (Nervous system disorders) | 11 (11)
Epilepsy (Nervous system disorders) | 7 (7)
Seizure cluster (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 2 (2)
Partial seizures with secondary generalisation (Nervous system disorders) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Cerebellar syndrome (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Cervical cord compression (Nervous system disorders) | 1 (1)
Complex partial seizures (Nervous system disorders) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1)
Encephalitis (Nervous system disorders) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Myelopathy (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1)
Simple partial seizures (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Suicide attempt (Psychiatric disorders) | 7 (7)
Suicidal ideation (Psychiatric disorders) | 5 (5)
Acute psychosis (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Aggression (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (3)
Delirium febrile (Psychiatric disorders) | 1 (1)
Emotional disorder (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1)
Spermatic cord haemorrhage (Reproductive system and breast disorders) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Intervertebral disc operation (Surgical and medical procedures) | 1 (1)
Tenodesis (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivaracetam (SS) (N=766)
Fatigue (General disorders) | 59 (67)
Nasopharyngitis (Infections and infestations) | 65 (102)
Upper respiratory tract infection (Infections and infestations) | 59 (101)
Urinary tract infection (Infections and infestations) | 57 (86)
Influenza (Infections and infestations) | 40 (47)
Contusion (Injury, poisoning and procedural complications) | 44 (71)
Fall (Injury, poisoning and procedural complications) | 43 (60)
Back pain (Musculoskeletal and connective tissue disorders) | 46 (59)
Arthralgia (Musculoskeletal and connective tissue disorders) | 41 (56)
Headache (Nervous system disorders) | 102 (187)
Dizziness (Nervous system disorders) | 100 (123)
Somnolence (Nervous system disorders) | 73 (88)
Depression (Psychiatric disorders) | 45 (53)
Anxiety (Psychiatric disorders) | 42 (48)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-05-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT01339559/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/59/NCT01339559/SAP_001.pdf